CLINICAL TRIAL: NCT02744924
Title: A Community-based Intervention to Increase Physical Activity Levels in Older Adults Using Citizen-science and Modern Technology
Brief Title: Intervention to Increase Physical Activity in Older Adults Using Citizen-science and Modern Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAPACITY
Record Dates: First submitted 2016-04-12; First posted 2016-04-20 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Sedentary; Elderly; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical activity intervention (Experimental): Participants undergo the community-based physical activity promotion (see Intervention)
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention — The intervention is comprised of 5 steps:
  1. Goal setting: Over a step-counter (smartphone app) participants learn about their daily average step count. They are coached to set individual goals
  2. Fitness assessment: To recommend suitable frequency and intensity of walking program using mapped trails
  3. Structured walking groups: Promoted and communicated via app. Participants can additionally organize walking groups of their own.
  4. Feedback: Participants will see individual and group data over the step-counter app, and they can communicate with others via a communication app. They will be incentivized to reach goals through a gamification approach.
  5. Invite friends: After 12 weeks, participants are encouraged to invite people who fulfil the inclusion criteria to join the project

SUMMARY:
To develop and implement a physical activity promotion intervention for older adults with or without chronic disease living in an urban environment.

DETAILED DESCRIPTION:
The World Health organization recommends that all adults should aim for 30 minutes of moderate physical activity on at least five days of the week. The importance of physical activity for promoting heath is complicated when considering inactive older adults and chronic conditions. A problematic cycle emerges where physical inactivity increases the likelihood for developing chronic conditions, and, in turn, many chronic conditions are associated with symptoms that make physical activity more difficult.

The investigators aim to develop and implement a physical activity promotion intervention for older adults with or without chronic disease living in an urban environment that considers individual, interpersonal and environmental factors and makes use of a citizen-science approach and modern PA-monitoring devices.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Living within or <5km from Wetzikon (Zurich area)
* Understand and speak German
* Number of repetitions in the 1-min sit-to-stand test below the 75th percentile compared to the Swiss population (age and sex-specific reference values)

Exclusion Criteria:

* Symptomatic / unstable cardiovascular disease
* Cardiac surgery within one year

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Physical activity as the average daily number of steps | Change from baseline to 6 months
  Average daily number of steps measured by accelerometry (Actigraph wGT3x) during 1 week

SECONDARY OUTCOMES:
Physical activity intensity | Change from baseline to 6 months
  Time spent in moderate-to-vigorous physical activity (min/day) measured by accelerometry (Actigraph wGT3x) during 1 week
Exercise capacity (1-minute sit-to-stand test) | Change from baseline to 6 months
  Number of repetitions performed in the 1-minute sit-to-stand test
Health-related quality of life | Change from baseline to 6 months
  Assessed by the EQ-5D
Symptoms of anxiety and depression | Change from baseline to 6 months
  Assessed by the Hospital Anxiety and Depression Scale
Health status | Change from baseline to 6 months
  Assessed by the Feeling Thermometer
Perceived social support | Change from baseline to 6 months
  Assessed by the short version of the Social Support Questionnaire

OTHER OUTCOMES:
Exploratory outcome: Course of daily number of steps | Daily number of steps during the intervention period (6 months)
  Exploration of course of number of steps measured by smartphone application
Exploratory outcome: Social connections | Through study completion, an average of 6 months
  Exploration of the use of the communication and calendar apps
Exploratory outcome: Participant satisfaction (questionnaire, quantitative) | Assessed at 6 months (follow-up)
  Assessed by self-administered questionnaire
Exploratory outcome: Participant satisfaction (interview, qualitative) | Assessed at 6 months (follow-up)
  Assessed by semi-structured interview
Safety outcome: Adverse events | Through study completion, an average of 6 months
  Adverse events are assessed, collected and reported according to guidelines
Physiological response to walking | At 1 day (during the intervention period)
  Physiological response during walking exercise using a metabolic cart in a subgroup of participants

CONTACTS AND LOCATIONS:
Overall Officials: Milo Puhan, Prof. Dr., Principal Investigator — EBPI, University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided